CLINICAL TRIAL: NCT02342366
Title: Multimodal Characterization of the Prosocial and Prosexual Effects of GHB Assessing Behavior, fMRI, EEG, and Neuroendocrine Mechanisms
Brief Title: Characterization of the Prosocial and Prosexual Effects of GHB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University of Regensburg (Other); University of Salerno (Other); University of Vienna (Other); University of Freiburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: PUK-GHB01
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Depressive Disorder, Major; Bipolar Disorder; Autistic Disorder
Keywords: Sodium Oxybate, Altruism, Neurostreroids, Liquid Ecstasy
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Autistic Disorder; Altruism | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: GHB 35 mg/kg p.o.; Drug: GHB 20 mg/kg p.o.
- GHB (Experimental): GHB, Gamma-Hydroxybutyrate, two doses (20 and 35 mg/kg p.o.)
  Interventions: Drug: GHB 35 mg/kg p.o.; Drug: GHB 20 mg/kg p.o.

INTERVENTIONS:
Drug: GHB 35 mg/kg p.o. — GHB 35 mg/kg p.o.
  Other Names: Sodium Oxybate
Drug: GHB 20 mg/kg p.o. — GHB 20 mg/kg p.o.
  Other Names: Sodium Oxybate

SUMMARY:
The purpose of this study is to determine whether gamma-Hydroxybutyrate (GHB) has prosocial and prosexual effects in healthy male participants, and to characterize these putative effects via behavioral tests, functional magnetic resonance imaging (fMRI), electroencephalography (EEG), and neuroendocrine parameters. The investigators predict that GHB in fact has prosocial and prosexual effects which can be neurobiologically characterized using the assessed methods. Such effects would be of high interest for the treatment of mental disorders which involve impairments of social interaction and sexual function such as major depression or autism.

DETAILED DESCRIPTION:
Introduction

Gammahydroxybutyrate (GHB) is an endogenous short-chain fatty acid and discussed as a neurotransmitter (Bessman and Fishbein, 1963) with high affinity to specific GHB (Benavides et al., 1982; Snead, 2000) and α4βδ-gamma-Aminobutyric acid (GABA)A receptors (Absalom et al., 2012) that also binds with lower affinity to GABAB receptors (Engberg and Nissbrandt, 1993). It is internationally used as standard treatment for narcolepsy with cataplexy (Alshaikh et al., 2012), and in some European countries for alcohol withdrawal and craving (Keating, 2014). Additionally, recent randomized controlled studies showed therapeutic effects in fibromyalgia (Spaeth et al., 2013). Anecdotal reports from GHB abusers indicate mood enhancing, prosocial and prosexual effects of the drug (Sumnall et al., 2008), which were not objectively assessed so far. Impaired social decision making is a behavioral finding in depression (Pulcu et al., 2014), that is related to social withdrawal symptoms. Moreover, sexual dysfunction is both a symptom of depression and an adverse effect of most antidepressant medications (Kennedy and Rizvi, 2009), with a deteriorating impact on quality of life measures. Due to its unique pharmacologic effects on sleep, daytime vigilance, pain, and social interaction, GHB was recently proposed as experimental therapeutic for the treatment of depression (Bosch et al., 2012).

Study Aims

A) Investigating the putative prosocial effects of GHB in humans B) Investigating the putative prosexual effects of GHB in humans C) Investigating the neuroendocrine mechanisms of putative prosocial and prosexual effects of GHB in humans D) Investigating electrophysiological effects of GHB in decision-making in humans E) Investigating the functional neurobiology of GHB and its putative prosexual effects in humans

Study Design

A) The effects of GHB on social cognition, sexual arousal, neuroendocrine parameters, and EEG measures in healthy subjects: GHB (20 mg/kg p.o.) was tested in 16 healthy males, using a randomized, placebo-controlled, cross-over design. Subjective effects on mood were assessed by visual analogue scales (VAS) and the GHB Specific Questionnaire (GSQ). Prosocial behavior was examined by the Charity Donation Task, the Social Value Orientation test, and the Reciprocity Task. We assessed reaction time and motor performance using the Delayed Matching to Sample and the Reaction Time tasks from the Cambridge Neuropsychological Test Automated Battery (CANTAB). We assessed social cognition using the Multifaceted Empathy Task (MET) and the Movie for the Assessment of Social Cognition (MASC). We assessed memory using a German version of the Rey Auditory Verbal Learing Task. Sexual arousal was assessed using the Sexual Arousal and Desire Inventory (SADI), sexual perception was assessed using a self-designed Sexual Arousal Task (SAT). Furthermore, the investigators assessed GHB effects on brain electrophysiological activity using electroencephalography (EEG) and a flanker task for the assessment of error-related negativity. Blood plasma levels of GHB, oxytocin, testosterone, progesterone, dehydroepiandrosterone (DHEA), cortisol, aldosterone, and adrenocorticotropic hormone (ACTH) were determined.

B) The effects of GHB on neuronal networks and sexual arousal in healthy subjects - an fMRI study: The investigators performed a characterization of the putative prosexual effects of GHB (35 mg/kg vs. placebo p.o.) in 19 healthy participants. Questionnaires (VAS, SADI, GSQ) were used to assess subjective aspects. Brain reactivity towards erotic vs. neutral pictures of persons, as well as resting state connectivity and arterial spin labelling (ASL) was investigated with functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects.

Exclusion Criteria:

* Any Axis-I DSM-IV psychiatric disorder, any form of addiction or regular illegal drug use (lifetime use >5 occasions) with exception of occasional cannabis use, a lifetime history of GHB use, a neurological disorder or head injury, clinically relevant medical diseases, a family history of schizophrenia or bipolar disorder, and any use of prescription drugs.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sexual Arousal | 14 days
  Changes in sexual arousal after GHB challenge compared to placebo (Sexual Arousal and Desire Inventory [SADI], Sexual Arousal Task [SAT], brain reactivity towards erotic vs. neutral pictures ([fMRI-Task])
Social Cognition and Behavior | 14 days
  Changes in social cognition and behavior after GHB challenge compared to placebo (Charity Donation Task, Social Value Orientation test, Reciprocity Task, Multifaceted Empathy Task [MET], Movie for the Assessment of Social Cognition [MASC])

SECONDARY OUTCOMES:
Composite measure of Neuroendocrine Parameters | 14 days
  Testosterone, DHEA, cortisol, aldosterone, ACTH, progesterone, oxytocin plasma levels after GHB challenge compared to placebo
electroencephalography (EEG) activity | 14 days
  EEG activity during a flanker task after GHB challenge compared to placebo
fMRI activity | 14 days
  Brain activity in fMRI after GHB challenge compared to placebo (Picture-Task, Resting State Connectivity, ASL)

CONTACTS AND LOCATIONS:
Overall Officials: Erich Seifritz, Professor, Principal Investigator — University of Zurich
Locations (1):
- Hospital for Psychiatry, University of Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Absalom N, Eghorn LF, Villumsen IS, Karim N, Bay T, Olsen JV, Knudsen GM, Brauner-Osborne H, Frolund B, Clausen RP, Chebib M, Wellendorph P. alpha4betadelta GABA(A) receptors are high-affinity targets for gamma-hydroxybutyric acid (GHB). Proc Natl Acad Sci U S A. 2012 Aug 14;109(33):13404-9. doi: 10.1073/pnas.1204376109. Epub 2012 Jul 2. PMID 22753476
- [Background] Alshaikh MK, Tricco AC, Tashkandi M, Mamdani M, Straus SE, BaHammam AS. Sodium oxybate for narcolepsy with cataplexy: systematic review and meta-analysis. J Clin Sleep Med. 2012 Aug 15;8(4):451-8. doi: 10.5664/jcsm.2048. PMID 22893778
- [Background] Benavides J, Rumigny JF, Bourguignon JJ, Cash C, Wermuth CG, Mandel P, Vincendon G, Maitre M. High affinity binding sites for gamma-hydroxybutyric acid in rat brain. Life Sci. 1982 Mar 15;30(11):953-61. doi: 10.1016/0024-3205(82)90624-5. PMID 7070203
- [Background] BESSMAN SP, FISHBEIN WN. GAMMA-HYDROXYBUTYRATE, A NORMAL BRAIN METABOLITE. Nature. 1963 Dec 21;200:1207-8. doi: 10.1038/2001207a0. No abstract available. PMID 14089913
- [Background] Bosch OG, Quednow BB, Seifritz E, Wetter TC. Reconsidering GHB: orphan drug or new model antidepressant? J Psychopharmacol. 2012 May;26(5):618-28. doi: 10.1177/0269881111421975. Epub 2011 Sep 17. PMID 21926421
- [Background] Engberg G, Nissbrandt H. gamma-Hydroxybutyric acid (GHBA) induces pacemaker activity and inhibition of substantia nigra dopamine neurons by activating GABAB-receptors. Naunyn Schmiedebergs Arch Pharmacol. 1993 Nov;348(5):491-7. doi: 10.1007/BF00173208. PMID 8114948
- [Background] Keating GM. Sodium oxybate: a review of its use in alcohol withdrawal syndrome and in the maintenance of abstinence in alcohol dependence. Clin Drug Investig. 2014 Jan;34(1):63-80. doi: 10.1007/s40261-013-0158-x. PMID 24307430
- [Background] Kennedy SH, Rizvi S. Sexual dysfunction, depression, and the impact of antidepressants. J Clin Psychopharmacol. 2009 Apr;29(2):157-64. doi: 10.1097/JCP.0b013e31819c76e9. PMID 19512977
- [Background] Pulcu E, Thomas EJ, Trotter PD, McFarquhar M, Juhasz G, Sahakian BJ, Deakin JF, Anderson IM, Zahn R, Elliott R. Social-economical decision making in current and remitted major depression. Psychol Med. 2015 Apr;45(6):1301-13. doi: 10.1017/S0033291714002414. Epub 2014 Oct 10. PMID 25300570
- [Background] Snead OC 3rd. Evidence for a G protein-coupled gamma-hydroxybutyric acid receptor. J Neurochem. 2000 Nov;75(5):1986-96. doi: 10.1046/j.1471-4159.2000.0751986.x. PMID 11032888
- [Background] Spaeth M, Alegre C, Perrot S, Wang Y, Guinta DR, Alvarez-Horine S, Russell I; Sodium Oxybate Fibromyalgia Study Group. Long-term tolerability and maintenance of therapeutic response to sodium oxybate in an open-label extension study in patients with fibromyalgia. Arthritis Res Ther. 2013 Nov 11;15(6):R185. doi: 10.1186/ar4375. PMID 24286114
- [Background] Sumnall HR, Woolfall K, Edwards S, Cole JC, Beynon CM. Use, function, and subjective experiences of gamma-hydroxybutyrate (GHB). Drug Alcohol Depend. 2008 Jan 1;92(1-3):286-90. doi: 10.1016/j.drugalcdep.2007.07.009. Epub 2007 Sep 4. PMID 17766059
- [Derived] Dornbierer DA, Boxler M, Voegel CD, Stucky B, Steuer AE, Binz TM, Baumgartner MR, Baur DM, Quednow BB, Kraemer T, Seifritz E, Landolt HP, Bosch OG. Nocturnal Gamma-Hydroxybutyrate Reduces Cortisol-Awakening Response and Morning Kynurenine Pathway Metabolites in Healthy Volunteers. Int J Neuropsychopharmacol. 2019 Oct 1;22(10):631-639. doi: 10.1093/ijnp/pyz047. PMID 31504554

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT02342366/Prot_SAP_000.pdf